#### 5. Appendices

# a. Appendix 1 (Information Sheet and Informed Consent)

"Effectiveness of the osteopathic treatment in patients with nonspecific cervical pain.

Randomized controlled pragmatic clinical trial "

#### Principal Investigators:

\* Óscar Hernandez (IntegroSalus), Edgar Segarra (Osteopatia Horta Clinic), David Puertas (Center Axis)

### Informational page

Dear Mr / Mrs:

The study in which we propose to participate, constitutes a scientific investigation in the field of cervical pain. This research is framed in the context of a final Master project. It is a study whose intervention does not generate any type of cost for the patient nor an increased risk in relation to the usual clinical practice, given that the interventions compared are common in osteopathic manual practice. The objective of this study is to compare the effect of 3 interventions. All of them have been shown to have positive effects in reducing cervical pain. Two of the interventions constitute different modalities of manual therapy, and the third is based on a specific exercise plan for cervical pain. If you agree to participate in this study, you will be required to complete two questionnaires related to cervical pain (50 questions) and quality of life (36 questions). The estimated time to complete the forms is 8 minutes and must be completed in three moments of the study (start, end of treatment, 1 month post-treatment). You will receive them by email again or you can fill them out electronically at any of the centers attached to the study

Participation is **VOLUNTARY**. At any time you can leave the study without giving any explanation. All personal data obtained in this study will be treated confidentially in accordance with the Organic Law of Protection of Personal Data 15/99 and the Regulation (EU) 2016/679 General Data Protection. The information obtained will be used exclusively for the specific purposes of this study, and will be coded to maintain the anonymity of the participants at all times.

Participants have the right to access, rectification, cancellation, opposition, to limit the processing of their data that are incorrect, to request a copy of them, or to transfer the data collected (portability) to a third party, and to exercise These rights must be communicated to the principal investigator.

In case of transfer of data to third countries outside the EU or the European Economic Area (EEA), the researcher will establish the necessary measures to guarantee a level of data protection equivalent to that granted by European legislation.

The research team will keep the records of this clinical study for a period of not less than 25 years.

\* This study project has been previously authorized by an independent Research Ethics Committee, which ensures respect for the rights, safety and well-being of people who participate in research projects.

| "Effectiveness of the osteopathic treatment in patients with nonspecific cervical pain. |
|---|
| Randomized controlled pragmatic clinical trial " |

| D 1 | | 1 | 45 | 4 |
|--------|-----|-------|------|-------|
| Princi | naı | inves | ะบดล | tors: |
| | ρα. | | 9 | |

\* Óscar Hernandez (IntegroSalus), Edgar Segarra (Osteopatia Horta Clinic), David Puertas (Center Axis)

# **Informed Consent**

We request your consent to participate in this study, which means that we can use the information obtained in the survey and record and analyze it later in the framework of this scientific research. Of course, if you do not participate in the study, in no case will this influence the professional care provided.

# PATIENT WRITTEN CONSENT

| | I, | , I read the sheet |
|---|---|---|
| | information that they have given me, I have been | n able to ask questions about the study, I have |
| received | enough information about it and I have been able | e to consult my doubts |
| | with Mr | |
| I understand that acceptance is voluntary and that I can leave the study whenever I want withougiving explanations, so I agree to participate in the study. | | |
| | Signature of the patient | Signature of the osteopath attending to him |